CLINICAL TRIAL: NCT05463068
Title: A Randomized, Observer-Blinded, Phase 3 Study to Compare the Immunogenicity and Safety of 3 Lots of NVX-CoV2373 in Adults
Brief Title: Study to Compare the Immunogenicity and Safety of 3 Lots of NVX-CoV2373 in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novavax (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019nCoV-307
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-07

CONDITIONS: COVID-19; SARS-CoV-2 Infection
Keywords: Coronavirus; COVID-19
MeSH Terms: conditions — COVID-19; Coronavirus Infections | interventions — NVX-CoV2373 adjuvated lipid nanoparticle

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Lot 1 (Experimental): 1 intramuscular (IM) injection of NVX-CoV2373 of 0.5 mL injection volume on Day 1.
  Interventions: Drug: NVX-Cov2373
- Lot 2 (Experimental): 1 intramuscular (IM) injection of NVX-CoV2373 of 0.5 mL injection volume on Day 1.
  Interventions: Drug: NVX-Cov2373
- Lot 3 (Experimental): 1 intramuscular (IM) injection of NVX-CoV2373 of 0.5 mL injection volume on Day 1.
  Interventions: Drug: NVX-Cov2373

INTERVENTIONS:
Drug: NVX-Cov2373 — Intramuscular (deltoid) injection of SARS-CoV-2 rS co-formulated with Matrix-M adjuvant (0.5 mL) on Day 1
  Other Names: SARS-CoV-2 rS/Matrix-M Adjuvant

SUMMARY:
This is a randomized, Phase 3 study comparing the immunogenicity and safety of 3 different lots of Novavax vaccine with Matrix-M™ adjuvant (NVX-CoV2373).The study will enroll approximately 900 previously vaccinated adults 18 to 49 years of age, inclusive.

DETAILED DESCRIPTION:
This is a randomized, Phase 3 study comparing the immunogenicity and safety of 3 different lots of Novavax vaccine with Matrix-M™ adjuvant (NVX-CoV2373). The study will enroll approximately 900 previously vaccinated adults 18 to 49 years of age, inclusive. Participants will be screened at baseline with the goal of enrolling approximately 900 previously vaccinated participants. Participants will be randomized 1:1:1 to receive 1 dose of the vaccine from 1 of 3 different lots, given on Day 1, at a dose level of 5 µg of antigen with 50 µg of Matrix-M adjuvant. All participants will remain on study for immunogenicity and safety data collection through 28 days following the vaccination.

ELIGIBILITY:
Inclusion Criteria:

To be included in this study, each individual must satisfy all of the following criteria:

1. Adults 18 to 49 years of age, inclusive, at screening
2. Willing and able to give informed consent prior to study enrollment and to comply with study procedures.
3. Participants of childbearing potential (defined as any participant who has experienced menarche and who is NOT surgically sterile [ie, hysterectomy, bilateral tubal ligation, or bilateral oophorectomy] or postmenopausal [defined as amenorrhea at least 12 consecutive months]) must agree to be heterosexually inactive from at least 28 days prior to enrollment and through the end of study (EOS) visit OR agree to consistently use a medically acceptable method of contraception from at least 28 days prior to enrollment and through the EOS visit.
4. Is medically stable, as determined by the investigator (based on review of health status, vital signs [to include body temperature], medical history, and targeted physical examination [to include body weight]). Vital signs must be within medically acceptable ranges prior to the study vaccination
5. Agree to not participate in any other SARS-CoV-2 prevention or treatment trials for the duration of the study.

   Note: For participants who become hospitalized with coronavirus disease 2019 (COVID-19), participation in investigational treatment studies is permitted.
6. Documented receipt of either 2 or 3 doses of the investigational Novavax vaccine with Matrix-M adjuvant (NVX- CoV2373); OR documented receipt of a full course of an FDA-authorized/approved COVID-19 vaccine; OR documented receipt of a full course of heterologous COVID-19 vaccines mentioned above. The most recent dose must have been administered at least 6 months prior to study vaccination.

Exclusion Criteria:

Participants meeting any of the following criteria will be excluded from the study.

1. History of laboratory-confirmed (by polymerase chain reaction [PCR] or rapid antigen test)COVID-19 infection ≤ 4 months prior to randomization.
2. Current participation in research involving receipt of an investigational product (drug/biologic/device).
3. Any known allergies or history of anaphylaxis to the active substance or any of the other ingredients contained in the investigational product.
4. Any autoimmune or immunodeficiency disease/condition (iatrogenic or congenital) or therapy that causes clinically significant immunosuppression.
5. Received any vaccine ≤ 90 days prior to study vaccination, except for influenza vaccine which may be received 4 days prior to study vaccine, or rabies vaccine which may be received at any time if medically indicated.
6. Received immunoglobulin, blood-derived products, or immunosuppressant drugs within 90 days prior to study vaccination, except for rabies immunoglobulin which may be given if medically indicated.
7. Active cancer (malignancy) on chemotherapy that is judged to cause significant immunocompromise within 1 year prior to first study vaccination (with the exception of malignancy cured via excision, at the discretion of the investigator).
8. Participants who are breastfeeding, pregnant, or who plan to become pregnant prior to the EOS visit.
9. Suspected or known history of alcohol abuse or drug addiction within 3 months prior to the study vaccine dose that, in the opinion of the investigator, might interfere with protocol compliance.
10. Any other condition that, in the opinion of the investigator, would pose a health risk to the participant if enrolled or could interfere with evaluation of the trial vaccine or interpretation of study results (including neurologic or psychiatric conditions likely to impair the quality of safety reporting).
11. Study team member or immediate family member of any study team member (inclusive of Sponsor, clinical research organization [CRO], and study site personnel involved in the conduct or planning of the study).
12. Participants with a history of myocarditis or pericarditis.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 911 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-08-17 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Serum Immunoglobulin G (IgG) Antibody Levels Expressed as GMEUs | Day 29
  IgG geometric mean ELISA unit concentrations (GMEU/mL) to the SARS-CoV-2 spike protein at Day 29 in each treatment arm.

SECONDARY OUTCOMES:
Serum IgG antibody levels expressed as seroconversion rate (SCR) | Day 29
  Proportion of participants in each treatment arm who achieve seroconversion (≥ 4-fold increase from baseline) in IgG concentrations to the SARS-CoV-2 spike protein at Day 29.
MN50 geometric mean titers (GMTs) to the SARS-CoV-2 expressed as GMTs | Day 29
  MN50 geometric mean titers to the SARS-CoV-2 spike protein at Day 29 in each treatment arm.
MN50 GMTs to the SARS-CoV-2 expressed as SCR | Day 29
  Proportion of participants in each treatment arm who achieve seroconversion (≥ 4-fold increase from baseline) in MN50 titers to the SARS-CoV-2 spike protein at Day 29.
Human Angiotensin-Converting Enzyme 2 (hACE2) inhibition assay titers GMT to the SARS-CoV-2 expressed as GMT | Day 29
  hACE2 inhibition assay titers (geometric mean titer [GMTs]) at Day 29 in each treatment arm.
hACE2 inhibition assay titers to the SARS-CoV-2 expressed as SCR | Day 29
  Proportion of participants in each treatment arm who achieve seroconversion (≥ 4-fold increase from baseline) in hACE2 titers concentrations to the SARS-CoV-2 spike protein at Day 29.
Incidence and severity of MAAEs | Day 0 to Day 29
  Incidence, duration, severity, and relationship of MAAEs through Day 29 (ie, 28 days after vaccine dose).
Incidence and severity of AESIs | Day 0 to Day 29
  Incidence, duration, severity, and relationship of AESIs (including myocarditis and/or pericarditis) through Day 29 (ie, 28 days after vaccine dose).
Incidence and relationship of SAEs | Day 0 to Day 29
  Incidence and relationship of SAEs throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Development, Study Director — Novavax, Inc.
Locations (30):
- United States (30):
  - Long Beach Clinical Trial Services Inc., Long Beach, California
  - Benchmark Research, Sacramento, California
  - Accel Clinical Research, DeLand, Florida
  - Research Centers of America, Hollywood, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Multi-Specialty Research Associates, Inc., Lake City, Florida
  - Cen/Excel ACMR, Atlanta, Georgia
  - Meridian Clinical Research, Savannah, Georgia
  - CRA Headlands, Stockbridge, Georgia
  - Velocity Clinical Research, Boise, Idaho
  - Meridian Clinical Research, Sioux City, Iowa
  - Meridian Clinical Research, Baton Rouge, Louisiana
  - MedPharmics, Gulfport, Mississippi
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research, Norfolk, Nebraska
  - Meridian Clinical Research, Omaha, Nebraska
  - Meridian Clinical Research, Endwell, New York
  - Rochester Clinical Research, Rochester, New York
  - OnSite Clinical Solutions, LLC, Charlotte, North Carolina
  - CTI Clinical Research Center, Cincinnati, Ohio
  - Velocity Clinical Research, Cleveland, Ohio
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Tekton Research, Yukon, Oklahoma
  - Velocity Clinical Research, Grants Pass, Oregon
  - Velocity Clinical Research, East Greenwich, Rhode Island
  - Benchmark Research, Austin, Texas
  - Tekton Research, Austin, Texas
  - Benchmark Research, Houston, Texas
  - Research Your Health, Plano, Texas
  - Tekton Research, San Antonio, Texas

REFERENCES:
- [Derived] Raiser F, Davis M, Adelglass J, Cai MR, Chau G, Cloney-Clark S, Eickhoff M, Kalkeri R, McKnight I, Plested J, Zhu M, Dunkle LM; 2019nCoV-307 study team. Immunogenicity and safety of NVX-CoV2373 as a booster: A phase 3 randomized clinical trial in adults. Vaccine. 2023 Sep 22;41(41):5965-5973. doi: 10.1016/j.vaccine.2023.07.056. Epub 2023 Aug 30. PMID 37652823